CLINICAL TRIAL: NCT01392469
Title: A Non-Randomized, Multiple Dose, Three Treatment Period, Open-Label, Single Sequence, Single Group Study to Evaluate the Pharmacokinetic Effect of Two Doses of QTI571 (Imatinib) on the Co-administered Drugs Sildenafil and Bosentan in Pulmonary Arterial Hypertension (PAH) Patients
Brief Title: Pharmacokinetic Effects of QTI571 on Sildenafil and Bosentan in Pulmonary Arterial Hypertension Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQTI571A2102; 2010-021344-17 (EudraCT Number)
Record Dates: First submitted 2011-05-10; First posted 2011-07-12 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary Vascular Resistance; Imatinib; Bosentan; Sildenafil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Imatinib Mesylate; Sildenafil Citrate; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib + Bosentan + Sildenafil (Experimental): Participants received treatment with bosentan 125 milligrams (mg) twice daily and sildenafil thrice daily for 8 days in treatment period 1. Participants were on the same sildenafil dose level (20, 40, 50 or 60 mg) they had been at study entry which was well tolerated in conjunction with bosentan. Following treatment period 1, the participants received concomitant treatment of oral imatinib 200 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 2. Following treatment period 2, the participants received concomitant treatment of oral imatinib 400 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 3.
  Interventions: Drug: Imatinib; Drug: Sildenafil; Drug: Bosentan

INTERVENTIONS:
Drug: Imatinib — Film coated tablets, oral administration
  Other Names: QTI571
Drug: Sildenafil — Oral Administration
Drug: Bosentan — Oral Administration

SUMMARY:
The purpose of this study was to investigate the effects of QTI571 (imatinib) on pharmacokinetics of bosentan and sildenafil at steady state when co-administered to participants with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Pulmonary arterial hypertension (PAH) in World Health Organization (WHO) Diagnostic Group 1, with pulmonary vascular resistance > 800 dyne*sec*cm^-5,
* On stable doses of bosentan and sildenafil

Exclusion Criteria:

* Other diagnosis of PAH in World Health Organization (WHO) Diagnostic Group 1 such as congenital large or small unrepaired systemic to pulmonary shunts, portal hypertension, Human Immunodeficiency Virus (HIV) infection, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic teleangiectasia, hemoglobinopathies, myeloproliferative disorders, veno-occlusive pulmonary disease
* Significant lung diseases not related to PAH
* Significant cardiovascular system disorders, hematological system disorders, liver insufficiency
* Significant diseases in other organ system.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04-20 (Actual); Primary Completion 2012-10-25 (Actual); Study Completion 2012-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (3):
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Weston, Florida
  - Novartis Investigative Site, Mineola, New York
- Novartis Investigative Site, Darlinghurst, New South Wales, Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Roma, RM, Italy
- Novartis Investigative Site, Vilnius, Lithuania
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with pulmonary arterial hypertension (PAH) were enrolled in the study at 8 investigation sites worldwide from 20 April 2011 to 25 October 2012.
Groups:
- Imatinib+ Bosentan+ Sildenafil: Participants received treatment with bosentan 125 mg twice daily and sildenafil thrice daily for 8 days in treatment period 1. Participants were on the same sildenafil dose level (20, 40, 50 or 60 mg) they had been at study entry which was well tolerated in conjunction with bosentan. Following treatment period 1, the participants received concomitant treatment of oral imatinib 200 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 2. Following treatment period 2, the participants received concomitant treatment of oral imatinib 400 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 3.
Period: Overall Study
Arm/Group | Imatinib+ Bosentan+ Sildenafil
Started | 21
Completed | 17
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled and who received at least one dose of study drug (bosentan, sildenafil, or imatinib).
Arm/Group | Imatinib+ Bosentan+ Sildenafil
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio of Dose Normalized Area Under the Curve From Time Zero to Tau (AUCtau) for Bosentan Before and After Imatinib Administrations
Description: AUCtau was the area under the curve calculated to the end of the dosing interval, tau. The effect of co-administration of imatinib at two doses (200 and 400 mg) on the pharmacokinetics of bosentan was performed on dose normalized AUCtau of bosentan. A mixed effects linear model was fitted to the log-transformed PK parameters. This model included treatment (i.e., dose of imatinib) as a fixed effect, and participant as a random effect. Estimates for the treatment differences and associated 90% confidence intervals were obtained from the above model. These estimates and confidence intervals were then "back-transformed" to the original scale, giving, for each dose level of imatinib, the ratio of imatinib + co-administered sildenafil and bosentan (test) relative to the co-administered drugs alone (sildenafil + bosentan) (reference).
Time Frame: Day 1: pre-dose, Day 8: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours post-dose, Day 9: pre-dose, Days 22 and 36: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Pharmacokinetics (PK) analysis set included all participants with data for at least one of the primary PK variables in at least one period and no major protocol deviations with impact on PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL/mg
Groups:
- Bosentan + Sildenafil (Reference): Participants received treatment with bosentan 125 mg twice daily and sildenafil thrice daily for 8 days in treatment period 1. Participants were on the same sildenafil dose level (20, 40, 50 or 60 mg) they had been at study entry which was well tolerated in conjunction with bosentan
- Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1): Following treatment period 1, the participants received concomitant treatment of oral imatinib 200 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 2.
- Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2): Following treatment period 2, the participants received concomitant treatment of oral imatinib 400 mg tablet daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 3.
Arm/Group | Bosentan + Sildenafil (Reference) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1) | Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2)
Number analyzed (Participants) | 17 | 17 | 17
hr*ng/mL/mg | 93.3 (49.9) | 109 (52.0) | 131 (38.0)
Statistical Analysis 1: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1); Test type: Superiority; Ratio (Test/Reference) = 1.17, 90% CI 2-sided [1.03 to 1.33]
Statistical Analysis 2: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2); Test type: Superiority; Ratio (Test/Reference) = 1.40, 90% CI 2-sided [1.23 to 1.59]

2. Primary Outcome: Geometric Mean Ratio of Dose Normalized AUCtau for Sildenafil Before and After Imatinib Administrations
Description: AUCtau was the area under the curve calculated to the end of the dosing interval, tau. The effect of co-administration of imatinib at two doses (200 and 400 mg) on the pharmacokinetics of sildenafil was performed on dose normalized AUCtau of sildenafil. A mixed effects linear model was fitted to the log-transformed PK parameters. This model included treatment (i.e., dose of imatinib) as a fixed effect, and participant as a random effect. Estimates for the treatment differences and associated 90% confidence intervals were obtained from the above model. These estimates and confidence intervals were then "back-transformed" to the original scale, giving, for each dose level of imatinib, the ratio of imatinib + co-administered sildenafil and bosentan (test) relative to the co-administered drugs alone (sildenafil + bosentan) (reference).
Time Frame: as for outcome 1
Population: PK analysis set included all participants with data for at least one of the primary PK variables in at least one period and no major protocol deviations with impact on PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL/mg
Arm/Group | Bosentan + Sildenafil (Reference) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1) | Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2)
Number analyzed (Participants) | 17 | 17 | 17
hr*ng/mL/mg | 7.22 (60.6) | 9.82 (42.5) | 12.3 (40.9)
Statistical Analysis 1: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1); Test type: Superiority; Ratio (Test/Reference) = 1.36, 90% CI 2-sided [1.14 to 1.62]
Statistical Analysis 2: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2); Test type: Superiority; Ratio (Test/Reference) = 1.70, 90% CI 2-sided [1.43 to 2.03]

3. Primary Outcome: Geometric Mean Ratio of Dose Normalized Maximum Plasma Concentration (Cmax) for Bosentan Before and After Imatinib Administrations
Description: Cmax was the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after dose administration. The effect of co-administration of imatinib at two doses (200 and 400 mg) on the pharmacokinetics of bosentan was performed on dose normalized Cmax of bosentan. A mixed effects linear model was fitted to the log-transformed PK parameters. This model included treatment (i.e., dose of imatinib) as a fixed effect, and participant as a random effect. Estimates for the treatment differences and associated 90% confidence intervals were obtained from the above model. These estimates and confidence intervals were then "back-transformed" to the original scale, giving, for each dose level of imatinib, the ratio of imatinib + co-administered sildenafil and bosentan (test) relative to the co-administered drugs alone (sildenafil + bosentan) (reference).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Bosentan + Sildenafil (Reference) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1) | Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2)
Number analyzed (Participants) | 17 | 17 | 17
ng/mL/mg | 21.9 (48.8) | 21.8 (60.3) | 23.4 (44.7)
Statistical Analysis 1: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1); Test type: Superiority; Ratio (Test/Reference) = 1.00, 90% CI 2-sided [0.82 to 1.21]
Statistical Analysis 2: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2); Test type: Superiority; Ratio (Test/Reference) = 1.07, 90% CI 2-sided [0.88 to 1.31]

4. Primary Outcome: Geometric Mean Ratio of Dose Normalized Cmax for Sildenafil Before and After Imatinib Administrations
Description: Cmax was the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after dose administration. The effect of co-administration of imatinib at two doses (200 and 400 mg) on the pharmacokinetics of sildenafil was performed on dose normalized Cmax of sildenafil. A mixed effects linear model was fitted to the log-transformed PK parameters. This model included treatment (i.e., dose of imatinib) as a fixed effect, and participant as a random effect. Estimates for the treatment differences and associated 90% confidence intervals were obtained from the above model. These estimates and confidence intervals was then "back-transformed" to the original scale, giving, for each dose level of imatinib, the ratio of imatinib + co-administered sildenafil and bosentan (test) relative to the co-administered drugs alone (sildenafil + bosentan) (reference).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Bosentan + Sildenafil (Reference) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1) | Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2)
Number analyzed (Participants) | 17 | 17 | 17
ng/mL/mg | 2.44 (68.6) | 3.14 (52.4) | 3.81 (52.9)
Statistical Analysis 1: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (200 mg/Day) + Bosentan + Sildenafil (Test 1); Test type: Superiority; Ratio (Test/Reference) = 1.28, 90% CI 2-sided [1.03 to 1.61]
Statistical Analysis 2: Comparison: Bosentan + Sildenafil (Reference) vs Imatinib (400 mg/Day) + Bosentan + Sildenafil (Test 2); Test type: Superiority; Ratio (Test/Reference) = 1.56, 90% CI 2-sided [1.24 to 1.95]

5. Secondary Outcome: Number of Participants With At Least One or More Adverse Events (AEs)
Description: An adverse event was the appearance or worsening of any undesirable sign, symptom, or medical condition that occurred after starting the study drug even if the event was not considered to be related to study drug. Number of participants with AEs were reported by treatment period.
Time Frame: From time of first administration of study drug until end of study (up to approximately 18 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Bosentan + Sildenafil: Participants received treatment with bosentan 125 mg twice daily and sildenafil thrice daily for 8 days in treatment period 1
- Imatinib (200 mg/Day) + Bosentan + Sildenafil: Following treatment period 1, the participants received concomitant treatment of oral imatinib 200 mg tablet daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 2.
- Imatinib (400 mg/Day) + Bosentan+ Sildenafil: Following treatment period 2, the participants received concomitant treatment of oral imatinib 400 mg tablet daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 3.
Arm/Group | Bosentan + Sildenafil | Imatinib (200 mg/Day) + Bosentan + Sildenafil | Imatinib (400 mg/Day) + Bosentan+ Sildenafil
Number analyzed (Participants) | 21 | 19 | 18
Participants | 10 | 9 | 16

6. Secondary Outcome: Dose Normalized Cmax of Imatinib and CGP74588 (Active Metabolite of Imatinib)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml/mg
Groups:
- Imatinib (200 mg/Day) + Bosentan + Sildenafil: Participants received concomitant treatment of oral imatinib 200 mg daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 2.
- Imatinib (400 mg/Day) + Bosentan + Sildenafil: Participants received concomitant treatment of oral imatinib 400 mg tablet daily, bosentan 125 mg twice daily and sildenafil thrice daily for 14 days in treatment period 3.
Arm/Group | Imatinib (200 mg/Day) + Bosentan + Sildenafil | Imatinib (400 mg/Day) + Bosentan + Sildenafil
Number analyzed (Participants) | 17 | 17
ng/ml/mg
  Imatinib Cmax/Dose | 7.55 (4.18) | 6.71 (3.39)
  CGP74588 Cmax/Dose | 1.37 (0.538) | 1.39 (0.575)

7. Secondary Outcome: Dose Normalized AUCtau of Imatinib and CGP74588 (Active Metabolite of Imatinib)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL/mg
Arm/Group | Imatinib (200 mg/Day) + Bosentan + Sildenafil | Imatinib (400 mg/Day) + Bosentan + Sildenafil
Number analyzed (Participants) | 17 | 17
hr*ng/mL/mg
  Imatinib AUCtau/Dose | 90.9 (49.3) | 88.4 (36.0)
  CGP74588 AUCtau/Dose | 19.3 (9.69) | 20.6 (9.07)

ADVERSE EVENTS:
Time Frame: From time of first administration of study drug until end of study (up to approximately 18 months)
Description: Safety analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement
Arm/Group | Bosentan + Sildenafil | Imatinib (200 mg/Day) + Bosentan + Sildenafil | Imatinib (400 mg/Day) + Bosentan+ Sildenafil | Total Participants
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/19 | 1/18 | 2/21
Other Adverse Events (participants affected / at risk) | 10/21 | 9/19 | 16/18 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan + Sildenafil (N=21) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (N=19) | Imatinib (400 mg/Day) + Bosentan+ Sildenafil (N=18) | Total Participants (N=21)
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan + Sildenafil (N=21) | Imatinib (200 mg/Day) + Bosentan + Sildenafil (N=19) | Imatinib (400 mg/Day) + Bosentan+ Sildenafil (N=18) | Total Participants (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 1 | 2
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 2 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4 | 2 | 7
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 5
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 3 | 5
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 3
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.